CLINICAL TRIAL: NCT07249242
Title: Healing Outcomes of Peri-implant Soft Tissues With Customized Healing Abutments in Immediate and Delayed Implant Placement Protocols: a Pilot Study
Brief Title: Healing Outcomes of Peri-implant Soft Tissues With Different Healing Abutments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006389
Record Dates: First submitted 2025-09-22; First posted 2025-11-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control: Pre Fabricated Healing Abutment (Active Comparator): Subjects that are randomized into the control group will have a pre-fabricated healing abutment used.
  Interventions: Device: Healing Abutment- pre fabricated
- Investigational: Customized Healing Abutment (Experimental): Subjects that are randomized into the control group will have a customized healing abutment used.
  Interventions: Device: Healing Abutment- customized

INTERVENTIONS:
Device: Healing Abutment- customized — A customized healing abutment will be used on subjects in this study as part of their implant healing process.
  Arms: Investigational: Customized Healing Abutment
Device: Healing Abutment- pre fabricated — A pre-fabricated (pre- made) healing abutment will be used on subjects in this study as part of their implant healing process.
  Arms: Control: Pre Fabricated Healing Abutment

SUMMARY:
The purpose of this study is to compare how well our research participants heal with two different kind of healing abutments used. One is pre-fabricated, meaning it is made to fit anyone, and the other is customized to fit the subject specifically. Much of what will occur is 'standard of care' meaning it is part of a subject's typical dental treatment and the research team wants to just look at the data for this research study, as well.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of record at TUSDM who are over 18 years of age
2. Implants placed as immediate or delayed with a torque of ≥ 35 Ncm eligible to receive a healing abutment left exposed to heal;
3. Site of implant placement not requiring soft tissue augmentation at the time of healing abutment placement
4. Sufficient mesial, distal space (7mm for anterior teeth and premolar and 8-9mm for molars) and interocclusal space (7-8mm for screw and cement retained crowns) for definitive restorations (12).

Exclusion Criteria:

1. Unable to give consent
2. active periodontal disease
3. Heavy smoker
4. Pregnant
5. Active infection at implant site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Soft tissue healing progress | 3 months
  Clinical Evaluation of Soft Tissue Healing; the clinician will perform intraoral examination on tissue color, contour, signs of inflammation, presence of keratinized tissue and soft tissue integration around the healing abutment. These are all visual observations and will be recorded as Yes/No.

SECONDARY OUTCOMES:
Functional outcome of gingival appearance | 3 months
  gingival appearance- reported through visual observation of presence of gingiva and color of implant and healing abutment. This observation is just on general healing progress related to this outcome, nothing is measured on a scale.
Functional outcome of implant esthetic | 3 months
  Implant esthetics - reported through visual observation of presence of gingiva and color of implant and healing abutment. This observation is just on general healing progress related to this outcome, nothing is measured on a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Mordini, Principal Investigator — Tufts University
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No